CLINICAL TRIAL: NCT02854423
Title: Long-term Comparison of Biodegradable Polymer Biolimus-eluting Stents and Durable-polymer Everolimus-eluting Stents in Patients With Diabetes Mellitus
Brief Title: Comparison of Biodegradable Polymer vs Durable-polymer in Diabetic Patients
Acronym: RUDI 2D
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gennaro Sardella, Professor, University of Roma La Sapienza
Other Study IDs: RUDI 2D
Record Dates: First submitted 2016-02-01; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Percutaneous Coronary Intervention; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- biodegradable polymer
  Interventions: Device: percutaneous coronary interventions
- durable-polymer
  Interventions: Device: percutaneous coronary interventions

INTERVENTIONS:
Device: percutaneous coronary interventions — Consecutive diabetic patients undergoing percutaneous coronary interventions with Biodegradable polymer Biolimus Eluting Stent or durable polymer Everolimus Eluting Stent implantation

SUMMARY:
Both biodegradable polymer-based biolimus-eluting stents (BP-BES) and durable polymer-based everolimus-eluting stents (DP-EES) have been shown to improve long-term clinical outcomes as compared with early generation DES. BP-BES with DP-EES have been directly compared in 2 randomized trials, showing no differences between the two devices in all-comer patients during long-term follow-up. It is unknown whether these results are consistent in real-world patients with diabetes mellitus during long-term follow-up. To evaluate the safety and efficacy profile of biodegradable polymer-coated biolimus-eluting stents (BP-BES) as compared to durable polymer-coated everolimus-eluting stents (DP-EES) in patients with diabetes mellitus during long-term follow-up.

Consecutive diabetic patients undergoing percutaneous coronary interventions with BP-BES or DP-EES implantation were included in a multicenter registry between January 2007 and May 2012. Long-term clinical outcomes between BP-BES and DP-EES will be compared using propensity score matching. The pre-specified primary endpoint is the occurrence of major cardiac adverse events (MACE) - a composite of all-cause death, myocardial infarction (MI) or target-vessel revascularization (TVR). Secondary endpoints are the individual components of the primary endpoint as well as definite stent thrombosis (ST).

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* diabetes mellitus
* percutaneous coronary interventions with biolimus eluting stent or everolimus eluting stent implantation
* signed informed consent

Exclusion Criteria:

* planned procedure requiring antiplatelet therapy withdrawal within 12 months from index coronary angioplasty
* patients with contraindication to dual antiplatelet therapy (aspirin plus ticlopidine or clopidogrel)
* known allergy to stent drugs

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive diabetic patients with coronary artery diseases undergoing percutaneous coronary interventions with BP-BES or DP-EES implantation between January 2007 and May 2012
Sampling Method: Probability Sample
Enrollment: 1347 (Actual)
Dates: Start 2007-01; Primary Completion 2012-05 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
major cardiac adverse events | 4 years
  a composite of all-cause death, myocardial infarction (MI) or target-vessel revascularization (TVR)

SECONDARY OUTCOMES:
rate of definite stent thrombosis in revascularized patients according with ARC definition | 4 years
Rate of composite of all-cause death in all participants | 4 years
Rate of myocardial infarction according with definition of MI type 1in all participants | 4 years
Rate of target-vessel revascularization (TVR) in all participants | 4 years